CLINICAL TRIAL: NCT03164824
Title: Thai Version of the Functional Rating Index for Patients With Back and Neck Pain: Cross-cultural Adaptation and Psychometric Properties Testing
Brief Title: Thai Version of Functional Rating Index
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: MahidolU_Wunpen3
Record Dates: First submitted 2017-01-08; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Questionnaire
Keywords: Questionnaire; Functional Rating Index; Cross-cultural adaptation; Psychometric properties testing
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaire — Cross-cultural adaptation stage:
  The FRI was cross-culturally adapted to Thai (called the Thai FRI) and the pre-final version of the Thai FRI was administered to patients.
  Psychometric properties testing stage:
  The questionnaires were administered 3 times: the first visit, the second visit and at 2 weeks.
  At the first visit: the patients with back pain completed the Thai FRI , Thai Roland-Morris Disability (Thai RM), Thai modified Oswestry Low Back Pain Disability (Thai modified ODQ), Thai multi-level Roland-Morris Disability (Thai multi-level RM). The patients with neck pain completed the Thai FRI and Thai Neck Disability Index.
  At the second visit: all patients completed the Thai FRI and Global Perceived Effect Scale (GPES).
  At 2 weeks: the patients completed the same questionnaires as the first visit. All patients and their treating physical therapists completed the GPES.

SUMMARY:
The purposes of this study were to conduct cross-cultural adaptation of the Functional Rating Index (FRI), to test psychometric properties of the translated questionnaire and to examine head-to-head comparisons with other questionnaires.

DETAILED DESCRIPTION:
This study comprised 2 major stages: 1) Cross-cultural adaptation and 2) psychometric properties testing.

Cross-cultural adaptation stage:

The FRI was cross-culturally adapted to Thai following the well-accepted guideline for the process of cross-cultural adaptation of self-report measure.

Psychometric properties testing stage:

The patients with back or neck pain completed the questionnaires at the first visit, the second visit and at 2-week (or at discharge or when reporting 80% improvement from the first visit).

ELIGIBILITY:
Inclusion Criteria

The participants were eligible if they were:

1. aged 18 years or older
2. seeking physical therapy treatment for a complaint of back and/or neck pain
3. able to understand, read, speak and write Thai

Exclusion Criteria:

The participants who were not willing to take part in the study, unable to understand, read, speak and write Thai were excluded from this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From physical therapy department in 9 settings in Thailand
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
questionnaire scores at the first visit | 20-25 minutes each time
  Back pain group: questionnaire scores from the Thai FRI, Thai RM, Thai modified ODQ, Thai multi-level RM; Neck pain group: questionnaire scores from the Thai FRI and Thai Neck Disability Index

SECONDARY OUTCOMES:
questionnaire scores at the second visit | 5 minutes each time
  questionnaire scores from the Thai FRI
Global Perceived Effect Scale (GPES) at the second visit | 3 minutes each time
  7-point GPES
questionnaire scores at 2 weeks | 20-25 minutes each time
  Back pain group: questionnaire scores from the Thai FRI, Thai RM, Thai modified ODQ, Thai multi-level RM; Neck pain group: Thai FRI, Thai Neck Disability Index
Global Perceived Effect Scale (GPES) at 2 weeks | 3 minutes each time
  7-point GPES

CONTACTS AND LOCATIONS:
Overall Officials: Wunpen Chansirinukor, PhD, Principal Investigator — Mahidol University

IPD SHARING:
Plan to Share IPD: No